CLINICAL TRIAL: NCT05622721
Title: Impact of Pet Contact on Antimicrobial-associated Dysbiosis and Clostridioides Difficile Infection
Brief Title: REMBRANDT: REcovery of the MicroBiome fRom Antibiotics for Dental implanTs
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Laurel Redding, Assistant Professor, University of Pennsylvania
Other Study IDs: 844131; 1K23AI163351-01A1 (NIH)
Record Dates: First submitted 2022-11-03; First posted 2022-11-21 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Dysbiosis; Clostridium Difficile; Pet-Human Bonding; Antibiotic-Associated Colitis
MeSH Terms: conditions — Dysbiosis; Human-Animal Bond; Enterocolitis, Pseudomembranous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pet owner: Pet owners
- Non pet owner: Non pet owners

SUMMARY:
Antimicrobial therapy can lead to disruption of the gut microbiome and infection with Clostridioides difficile, a disease associated with high morbidity and mortality, particularly among the elderly. Drawing on observations that pet ownership and close contact with pets are protective against colonization with C. difficile and recurrence of C. difficile infection, the proposed study will test the hypothesis that microbiota that provide colonization resistance against C. difficile are shared between patients and their pets and that pet contact can mitigate antimicrobial-associated gut dysbiosis and the risk of C. difficile infection. This study will further define epidemiologic and pathophysiologic characteristics of C. difficile infection and gut microbiome dysbiosis that could enhance therapeutic options for these conditions, potentially through non-invasive interventions involving animal contact.

DETAILED DESCRIPTION:
Clostridioides difficile infection (CDI) is one of the most common causes of healthcare-associated infectious diarrhea and results in significant morbidity and mortality. CDI occurs when the native gut microbiome is disrupted, most often following antimicrobial therapy, and the consequent dysbiosis results in a decrease in microbial diversity, changes in abundance of certain bacterial taxa, and loss of colonization resistance against C. difficile. Restoration of a "functionally intact" gut microbiome is critical to clearing C. difficile, and inadequate restoration can lead to recurrent CDI. The recovery of the gut microbiome from dysbiosis is poorly understood, and factors associated with having and re-gaining a providing colonization resistance against C. difficile are not well known. While animal reservoirs can serve as potential sources of pathogenic bacteria, studies by the candidate and other investigators found that pet ownership protects against colonization and re-infection with C. difficile. Moreover, microbiota are shared between pets and their owners, and the microbiomes of pets contain bacterial taxa that provide colonization resistance against C. difficile. Based on these data, the proposed research will 1) test the hypothesis that the observed protective effects of pet ownership are due to sharing of microbiota that provide colonization resistance against C. difficile between pets and owners; 2) determine whether pet contact mitigates antimicrobial-associated disruption of the gut microbiome and enhances its recovery; and 3) assess whether pet contact decreases the likelihood of colonization and infection with C. difficile following antimicrobial therapy. This will be accomplished though longitudinal sampling of the gut microbiome within the patient/pet unit among patients receiving prophylactic antimicrobials for non-enteric indications (dental implants).

The study will further define epidemiologic and pathophysiologic characteristics of CDI that could enhance therapeutic options for this disease. The underlying premise that animals are a source of protective microbiota rather than a reservoir of C. difficile represents a paradigm shift in CDI epidemiology that may identify animal contact as a novel microbiome-based form of therapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Receiving a dental implant.
* Ability to understand study procedures and to comply with them for the entire length of the study.

Exclusion Criteria:

* Antimicrobial therapy or hospitalization in the prior three months;
* Any gastrointestinal illness or underlying pathology (e.g., Inflammatory Bowel Disease, gastric ulceration)
* Sustained diarrheal disease (i.e., at least 3 episodes of loose or watery stool per day for 3 or more days) in the prior 3 months;
* Prior history of CDI in the prior year;
* Immunomodulating medication (e.g., tumor necrosis factor inhibitors or systemic steroids) or conditions (e.g., leukemia)
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source population will include patients over 18 years of age receiving prophylactic oral antimicrobials for dental implants at the University of Pennsylvania School of Dental Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Longitudinal change in diversity and composition of the gut microbiota following oral antibiotic prophylaxis | 90 days
  Changes in alpha diversity, beta diversity and composition of the gut microbiome will be ascertained between baseline (prior to taking antibiotics) and 3, 10, 30 and 90 days following the start of the antibiotic regimen
Colonization or infection with C. difficile following antibiotic prophylaxis | 3 days
  The presence of C. difficile in patients' stool will be determined before and 3 days after the beginning of the antibiotic regimen

CONTACTS AND LOCATIONS:
Overall Officials: Laurel Redding, VMD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- The Robert Schattner Center, University of Pennsylvania, School of Dental Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Any data, specimens, forms, reports, video recordings, and other records that leave the site will be identified only by a participant identification number (Participant ID, PID) to maintain confidentiality. All records will be kept in a locked file cabinet. All computer entry and networking programs will be done using PIDs only. Information will not be released without written permission of the participant, except as necessary for monitoring by the IRB or NIAID.
  Any presentation, abstract, or manuscript will be made available for review by the sponsor and the NIAID prior to submission.

DOCUMENTS (2):
  • Statistical Analysis Plan (2022-11-03): https://cdn.clinicaltrials.gov/large-docs/21/NCT05622721/SAP_000.pdf
  • Informed Consent Form (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/21/NCT05622721/ICF_001.pdf